CLINICAL TRIAL: NCT03866863
Title: Intra Uterine Growth Restriction. Minimum Required Evidence-based Care and Neonatal Prognosis: Impact of Healthcare Pathways
Brief Title: Intra Uterine Growth Restriction
Acronym: IUGR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: IUGR
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HFME births.: All birth more than 24 + 0 weeks of amenorrhea at the maternity ward of the hospital Femme-Mère-Enfant from 1st of january 2011 to 31 december 2017.
  Interventions: Other: Intrauterine growth restriction (IUGR)

INTERVENTIONS:
Other: Intrauterine growth restriction (IUGR) — Collection of number of patient's diagnosed with IUGR as defined in accordance with the consensus-based definition for early and late IUGR : birthweight < 3rd centile using French AUDIPOG curves adjusted for term and sex or estimated fetal weight < 10th centile combined with umbilical artery pulsatility index > 95th centile or breakage of growth.

SUMMARY:
Intrauterine growth restriction (IUGR) is associated with an increase in perinatal mortality and morbidity, as well as longer-term neurological, cognitive, cardiovascular and endocrine complications. In Europe, about 400,000 pregnancies per year are complicated by IUGR. However, antenatal diagnosis seems insufficient in clinical practice, making it impossible to recognize up to 75% of foetuses with IUGR. At a time when the use of good clinical practice has demonstrated a significant improvement in neonatal survival without severe morbidity, foetuses with IUGR are less likely to receive optimal care. Our hypothesis is that the rate of IUGR diagnosed underestimates the rate of actual IUGR.

ELIGIBILITY:
Inclusion Criteria:

* All birth more than 24 + 0 weeks of amenorrhea at the maternity ward of the hospital Femme-Mère-Enfant
* from 1st of january 2011 to 31 december 2017.

Exclusion Criteria:

* Infants born out of the hospital and secondarily hospitalized in the hospital Femme-Mère-Enfant .
* Multiple pregnancies,
* children with congenital fetal anomalies
* pregnancies without first trimester ultrasound (to date the pregnancy)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All birth more than 24 + 0 weeks of amenorrhea at the maternity ward of the hospital Femme-Mère-Enfant from 1st of january 2011 to 31 december 2017.
Sampling Method: Non-Probability Sample
Enrollment: 31052 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients diagnosed with Intrauterine growth restriction | Between 2011 and 2017
  IUGR was defined in accordance with the consensus-based definition for early and late IUGR : birthweight < 3rd centile using French AUDIPOG curves adjusted for term and sex or estimated fetal weight < 10th centile combined with umbilical artery pulsatility index > 95th centile or breakage of growth.

CONTACTS AND LOCATIONS:
Overall Officials: Muriel DORET, Prof., Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France